CLINICAL TRIAL: NCT03278977
Title: Apparent Life Threatening Events, Sudden Infant Death Syndrome and Muscarinic Receptors
Acronym: iALTE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Groupement Interrégional de Recherche Clinique et d'Innovation Est (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 6432
Record Dates: First submitted 2017-08-31; First posted 2017-09-12 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Apparent Life-Threatening Event in Infants Under One Year of Age
Keywords: Apparent Life-Threatening Event; ALTE; Sudden Infant Death
MeSH Terms: conditions — Brief, Resolved, Unexplained Event; Sudden Infant Death | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blood sample analysis will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALTE group (Other): Infants aged between 28 days and 12 months presenting severe(s) syncope(s) requiring hospitalization, for which a cause was identified during hospitalization.
  Interventions: Biological: Blood sample for specific analyzes
- iALTE group (Other): Infant aged between 28 days and 12 months presenting a severe syncope(s) requiring hospitalization, for which no etiology was found during hospitalization.
  Interventions: Biological: Blood sample for specific analyzes

INTERVENTIONS:
Biological: Blood sample for specific analyzes — Standard management of ALTE
  * Hospitalization in pediatric intensive care unit or pediatric emergencies
  * Etiologic research
  * Blood volume, 2.5mL in PaxGene® tube, for specific analyzes (M2R, AchE)

SUMMARY:
Apparent Life-Threatening Events (ALTE) in infants often lead to severe neurological complications or to sudden death. In such situations, cardio-pediatricians and intensive care physicians have no specific diagnosis or treatment. In a recent translational research (INSERM-DHOS), our team has reported a myocardiac abnormality in a rabbit model of vagal hyperreactivity which is also present in the human hearts of infants deceased from sudden death, i.e. increased M2 muscarinic receptors (M2R) density associated with compensative increased enzymatic activity and overexpression of acetylcholine esterase (AchE). In a recent PHRC-I study (article in preparation), these abnormalities have also been observed in the blood of patients, infants as well as adults, exhibiting severe vagal syncopes. We observed, even more importantly, similar abnormalities in infants under 1 year of age with very severe idiopathic ALTE (iALTE) compared with normal subjects and with patients who presented ALTE with identified etiologies (JAMA Pediatric, 2016 May). The aim of this present study is to validate the overexpression of M2R as a marker of risk of iALTE in infant under 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Infant aged between 28 days and 12 months, presenting severe syncope(s) requiring medical management, hospitalized in a pediatric intensive care unit or pediatric emergencies
* Consent signed and dated by the legal representatives
* Patients affiliated to a social security system

Exclusion Criteria:

* Infant with known cardiovascular, neurologic, infectious, toxic or metabolic pathologies before enrollment (before the syncope)
* Subject on medication for more than 3 months before enrollment
* Impossibility to clearly inform the legal representatives (comprehension problems)
* Subject in exclusion period for clinical trial (previous or current study)

Ages: 28 Days to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2018-09-15 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Muscarinic M2 receptor mRNA expression in blood | At the admission in the hospital, within 24 hours after the inclusion in the study
  Blood sample will be collected not later than 24 hours after the inclusion in the study and will be frozen until centralized analysis.
  A qRT-PCR will be performed for quantification of CHRM2 gene expression in blood (mRNA expression).
  Interim analysis with the 7-8 first samples per group together. Final analysis with all samples at the study completion.

SECONDARY OUTCOMES:
Acetylcholinesterase mRNA expression in blood | At the admission in the hospital, within 24 hours after the inclusion in the study.
  Blood sample will be collected not later than 24 hours after the inclusion in the study and will be frozen until centralized analysis..
  A qRT-PCR will be performed for quantification of ACHE gene expression in blood (mRNA expression).
  Interim analysis with the 7-8 first samples per group together. Final analysis with all samples at the study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Charlie DE MELO, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (4):
- France (4):
  - Pediatric Intensive Care unit/Emergency unit - Besançon University Hospital, Besançon
  - Pediatric Intensive Care Unit - Brabois Hospital - Nancy University Hospital, Nancy
  - Pediatric unit - Maison Blanche Hospital - Reims University Hospital, Reims
  - Pediatric intensive care unit/ Pediatric unit- Strasbourg University Hospital - Hautepierre Hospital, Strasbourg

IPD SHARING:
Plan to Share IPD: No